CLINICAL TRIAL: NCT05999474
Title: Combined Fractional CO2 Laser With Topical Tioconazole Versus Q-switched Nd:YAG Laser in the Treatment of Onychomycosis; a Randomized Controlled Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Elbendary, Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kasr Alainy
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Onychomycosis of Fingernail
MeSH Terms: interventions — tioconazole; Lasers

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional CO2 laser combined with topical tioconazole (Experimental): Fractional CO2 laser (10,600 nm) will be done. The sessions will be done every 2 weeks.
  Topical tioconazole 28% nail solution will be applied in between the sessions twice daily
  Interventions: Drug: Topical tioconazole
- Q switched ND-Yag (Active Comparator): Laser protocol with a specific parameters will be applied on the affected nails. In one session two passes across each nail plate will be performed with two minutes pauses between each pass. Sessions will be done every 2 weeks
  Interventions: Drug: Topical tioconazole

INTERVENTIONS:
Drug: Topical tioconazole — Laser
  Other Names: Laser

SUMMARY:
Our aim is to assess the clinical efficacy and the safety of fractional CO2 laser combined with topical tioconazole versus Q-switched Nd:YAG laser in the treatment of OM.

ELIGIBILITY:
Inclusion Criteria:

* • Age group >18 years.

  * Patients of both genders.
  * Patients with OM any type.

Exclusion Criteria:

* • Pregnancy

  * Localized bacterial infection around the affected nail
  * Concomitant nails disease that causes nail dystrophy or discoloration such as psoriasis, lichen planus and atopic dermatitis that may interfere with diagnosis and treatment
  * Hypersensitivity to terbinafine
  * Intake of oral antifungal medication within the last 3 months or used topical antifungal medication within the last 2 weeks prior to the laser treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
treatment of onychomycosis | 6 months
  Patient Evaluation (Clinical percentage of improvement). 2- Improvement of OM (assessed by investigator). 3-Percentage of grading and OSI score improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No